CLINICAL TRIAL: NCT01225237
Title: Post-marketing Clinical Study of Ramosetron Hydrochloride (Irribow Tablets) - Double-blind, Parallel-group Comparative Study in Patients (Male) With Diarrhea-predominant Irritable Bowel Syndrome
Brief Title: A Study to Evaluate Efficacy of Ramosetron on Diarrhea-predominant Irritable Bowel Syndrome (IBS) in Male Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 060-CL-501
Record Dates: First submitted 2010-10-19; First posted 2010-10-20 (Estimated); Last update posted 2014-10-15 (Estimated); Status verified 2014-10

CONDITIONS: Irritable Bowel Syndrome
Keywords: diarrhea; IBS; Colonic disease; YM060
MeSH Terms: conditions — Irritable Bowel Syndrome; Diarrhea; Colonic Diseases | interventions — ramosetron

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ramosetron group (Experimental)
  Interventions: Drug: Ramosetron
- Placebo group (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ramosetron — oral
  Other Names: Irribow; YM060
  Arms: ramosetron group
Drug: Placebo — oral
  Arms: Placebo group

SUMMARY:
A study to verify the superiority of ramosetron hydrochloride (Irribow Tablets) to placebo for male patients with diarrhea-predominant irritable bowel syndrome (D-IBS) and to evaluate its safety.

ELIGIBILITY:
Inclusion Criteria:

* Patients meeting the Rome III Diagnostic Criteria
* Loose (mushy) or watery stools within the last 3 months

Exclusion Criteria:

* Patients with a history of surgical resection of the stomach, small intestine or large intestine
* Patients with a history or current diagnosis of inflammatory bowel disease (Crohn's disease or colitis ulcerative)
* Patients with a history or current diagnosis of colitis ischemic
* Patients with a current diagnosis of enteritis infectious
* Patients with a current diagnosis of hyperthyroidism or hypothyroidism
* Patients who are currently participating in another clinical trial (including a post-marketing clinical study) or those who participated in another clinical trial (including a post-marketing clinical study) within 12 weeks before the study
* Patients with a history or current diagnosis of malignant tumor
* Patients with a history of abuse of drugs or alcohol within 1 year or those who are currently abusing them

Ages: 20 Years to 64 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 296 (Actual)
Dates: Start 2010-10; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Responder rate of stool form normalization | For 4 weeks

SECONDARY OUTCOMES:
Responder rate of patients reported global assessment of relief of IBS symptoms | For 4 weeks
Responder rate of patients reported assessment of relief of abdominal discomfort and/or pain | For 4 weeks
Responder rate of patients reported assessment of improvement of abnormal bowel habits | For 4 weeks
Safety assessed by the incidence of adverse events and abnormal values in labo-tests | For 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Chair — Astellas Pharma Inc
Locations (4):
- Japan (4):
  - Hokkaido
  - Kansai
  - Kantou
  - Kyusyu

REFERENCES:
- [Background] Fukudo S, Ida M, Akiho H, Nakashima Y, Matsueda K. Effect of ramosetron on stool consistency in male patients with irritable bowel syndrome with diarrhea. Clin Gastroenterol Hepatol. 2014 Jun;12(6):953-9.e4. doi: 10.1016/j.cgh.2013.11.024. Epub 2013 Dec 4. PMID 24315882